CLINICAL TRIAL: NCT02191124
Title: Measurement-based Care vs. Standard Care for Major Depressive Disorder: a Randomized Controlled Trial With Masked Raters
Brief Title: The Measurement-based Care in Patients With Depressive Disorder: A Randomized Controlled Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Gang Wang, vice-director of Affective Disorder Center, Beijing Anding Hospital, Capital Medical University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 2009-1051
Record Dates: First submitted 2014-07-10; First posted 2014-07-16 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Major Depressive Disorder
Keywords: Measurement-based care; Unipolar depression; Outpatients
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder | interventions — Paroxetine; Mirtazapine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- measurement-based care (Experimental): MBC allows psychiatrists to individualize treatment decisions for each patient based on the change of psychopathology and tolerance toward antidepressants. Treatment decisions were made by treating psychiatrists according to ratings of self-report scales obtained at each treatment visit. Paroxetine was started at 20mg/day and then raised to 30mg/day by week 4, 40mg/day by week 6, 50mg/day by week 8 and 60mg/day by week 10. Mirtazapine was started at 15mg/day and raised to 30mg/day by week 1 and 45mg/day by week 4. Dose adjustments were dependent on how long a patient had received a particular dose, symptom changes and side effects.
  Interventions: Drug: Paroxetine; Drug: Mirtazapine
- Standard treatment (Active Comparator): Patients in the ST group are treated by their psychiatrists according to their clinical needs as judged at each outpatient visit, receiving either open-label paroxetine (20-60mg/day) or mirtazapine (15-45mg/day) within the therapeutic dose range.
  Interventions: Drug: Paroxetine; Drug: Mirtazapine

INTERVENTIONS:
Drug: Paroxetine — Patients in both groups (MBC or ST) receive open-label paroxetine (20-60mg/day) within the therapeutic dose range recommended by the Guidelines for the Prevention and Treatment of Major Depression in China.
  Other Names: Seroxat
Drug: Mirtazapine — Patients in both groups (MBC or ST) receive open-label mirtazapine (15-45mg/day) within the therapeutic dose range recommended by the Guidelines for the Prevention and Treatment of Major Depression in China
  Other Names: Remeron

SUMMARY:
In recent years, measurement-based care (MBC) has been gaining more attention in the treatment of depression because it allows psychiatrists to individualize treatment decisions for each patient based on the change of psychopathology and tolerance toward antidepressants. Several studies, such as the Sequenced Treatment Alternatives to Relieve Depression (STAR*D) trial using MBC, found that MBC-informed sequential algorithms can be successfully integrated into clinical practice and improve patients' outcomes However, despite a strong theoretical rationale for MBC and data supporting the ability to implement MBC in clinical practice settings, there is currently no randomized controlled trial in MDD patients comparing MBC with usual/standard care. The investigators compare MBC with clinician's treatment decisions, standardizing care to two commonly prescribed antidepressants.

Therefore, the aim of this study is to determine the effects of MBC in patients with MDD compared to standard treatment (ST). The research hypothesis is that compared to ST, the estimated time to response and to remission would be significantly shorter in the MBC group without increased dropout rates and side effect burden.

DETAILED DESCRIPTION:
Objective: To compare the effectiveness and feasibility of the measurement-based care (MBC) in the treatment of depression with clinician's treatment decisions, standardizing treatment (ST, clinicians' choice decisions) to two commonly prescribed antidepressants.

Methods: Selecting the patients in psychiatric hospitals and general hospitals with depression, with multi-center randomized controlled study design. Refer to STAR-D "measurement-based care" mode, to establish the whole measurement-based evaluation system. Eligible patients will be randomly assigned to 24 weeks of MBC or ST, restricting treatment to paroxetine (20-60mg/day) or mirtazapine (15-45mg/day) in both groups. the ST group will maximize simulate of the actual clinical situation, and the patients of the MBC group are required to complete the prospective Life-chart Methodology (LCM-p), 16-item Quick Inventory of Depressive Symptomatology Self-Report (QIDS-SR16) and other related symptoms and side effects of self-assessment, the doctor will make a comprehensive assessment according to the results of self-assessment, adjust treatment according to research programs. This is 1-year follow-up study; the independent members will have a blinded assessment in the baseline visit and each point of view. Depressive symptoms are measured using the Hamilton Rating Scale for Depression (HAMD) and QIDS-SR.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-65 years;
2. outpatients;
3. diagnosis of non-psychotic MDD established by treating psychiatrists and confirmed by a checklist based on DSM-IV criteria at study entry ;
4. total score of HAMD-17≥17;
5. ability to communicate and provide written consent.

Exclusion Criteria:

1. current or past history of drug and alcohol dependence, bipolar, psychotic, obsessive-compulsive, or eating disorders;
2. history of lack of response or intolerance to any of the two protocol antidepressants (paroxetine or mirtazapine);
3. being pregnant or breast-feeding;
4. suicide attempts in the current depressive episode or major medical conditions contraindicating the use of the protocol antidepressants.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2011-06; Primary Completion 2012-11 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
The estimated time from randomization to response and remission according to Hamilton Rating Scale for Depression (HAMD) total score. | From randomization to response and remission (24 week))
  Response was defined as ≥50% decrease in the baseline HAMD total score; remission was defined as the HAMD total score ≤7

SECONDARY OUTCOMES:
The changes of Hamilton Rating Scale for Depression (HAMD) total score | From randomization to endpoint (Week 24)
  To measure the change of the severity of depressive symptoms
The incidence and nature of overall adverse events | From enrollment to endpoint (Week 24)
The incidence and nature of drug-related adverse events | From enrollment to endpoint (Week 24)
The number of subject withdrawal due to adverse events during double-blind phase | From randomization to endpoint(Week 24)
The changes of Quick Inventory of Depressive Symptomatology-Self-Report (QIDS-SR) total score | From randomization to endpoint (Week 24)
The changes of Frequency, Intensity, and Burden of Side Effects-Rating (FIBSER) | From randomization to endpoint (Week 24)
  The FIBSER is a self-report instrument assessing three domains of medication side effects within the past week

CONTACTS AND LOCATIONS:
Overall Officials: Gang Wang, MD;PhD, Principal Investigator — Beijing Anding Hospital, Capital Medical University
Locations (1):
- Beijing Anding Hospital, Beijing, Beijing Municipality, China